CLINICAL TRIAL: NCT01037309
Title: A Phase I/IIa, Open Label, Escalating Dose, Pilot Study to Assess the Effect, Safety, Tolerability and Pharmacokinetics of Multiple Subcutaneous and Intravenous Doses of PRO044 in Patients With Duchenne Muscular Dystrophy
Brief Title: Phase I/II Study of PRO044 in Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO044-CLIN-01
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PRO044, cohort 1 (Experimental): Subcutaneous injection of 0.5 mg/kg on day 1, 8, 15, 22 and 29.
  Interventions: Drug: PRO044 SC
- PRO044, cohort 2 (Experimental): Subcutaneous injection of maximally 1.5 mg/kg on day 1, 8, 15, 22 and 29.
  Interventions: Drug: PRO044 SC
- PRO044, cohort 3 (Experimental): Subcutaneous injection of maximally 5 mg/kg on day 1, 8, 15, 22 and 29.
  Interventions: Drug: PRO044 SC
- PRO044, cohort 4 (Experimental): Subcutaneous injection of maximally 8 mg/kg on day 1, 8, 15, 22 and 29.
  Interventions: Drug: PRO044 SC
- PRO044, cohort 5 (Experimental): Subcutaneous injection of maximally 10 mg/kg on day 1, 8, 15, 22 and 29
  Interventions: Drug: PRO044 SC
- PRO044, cohort 6 (Experimental): Subcutaneous injection of maximally 12 mg/kg on day 1, 8, 15, 22 and 29
  Interventions: Drug: PRO044 SC
- PRO044, cohort 7 (Experimental): Intravenous injection of maximally 1.5 mg/kg on day 1, 8, 15, 22 and 29
  Interventions: Drug: PRO044 IV
- PRO044, cohort 8 (Experimental): Intravenous injection of maximally 5 mg/kg on day 1, 8, 15, 22 and 29
  Interventions: Drug: PRO044 IV
- PRO044, cohort 9 (Experimental): Intravenous injection of maximally 8 mg/kg on day 1, 8, 15, 22 and 29
  Interventions: Drug: PRO044 IV

INTERVENTIONS:
Drug: PRO044 SC — Subcutaneous injection, once a week, for five weeks
  Arms: PRO044, cohort 1; PRO044, cohort 2; PRO044, cohort 3; PRO044, cohort 4; PRO044, cohort 5; PRO044, cohort 6
Drug: PRO044 IV — Intravenous injection, once a week, for five weeks
  Arms: PRO044, cohort 7; PRO044, cohort 8; PRO044, cohort 9

SUMMARY:
The purpose of this study is to see whether PRO044 is safe and effective to use as medication for DMD patients with a mutation around location 44 in the DNA for the dystrophin protein.

DETAILED DESCRIPTION:
To assess the effect of PRO044 at different dose levels in subjects with Duchenne muscular dystrophy To assess the safety and tolerability of PRO044 at different dose levels in subjects with Duchenne muscular dystrophy To determine the pharmacokinetics of PRO044 at different dose levels after subcutaneous and intravenous administration in subjects with Duchenne muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Boys aged between 5 and 16 years inclusive.
2. Duchenne muscular dystrophy resulting from a mutation correctable by treatment with PRO044.
3. Life expectancy of at least 6 months.
4. No previous treatment with investigational medicinal treatment within 6 months prior to the start of the (pre)-screening for the study.
5. No previous treatment with idebenone within 6 months prior to the start of the (pre)-screening for the study.
6. Willing and able to adhere to the study visit schedule and other protocol requirements.
7. Written informed consent signed (by parent(s)/legal guardian and/or the patient, according to the local regulations).
8. Glucocorticosteroids use which is stable for at least 2 months prior first drug administration.

Exclusion Criteria:

1. Aberrant RNA splicing and/or aberrant response to PRO044, detected by in vitro PRO044 assay during pre-screening.
2. Known presence of dystrophin in ≥ 5% of fibers in a pre-study diagnostic muscle biopsy.
3. Severe muscle abnormalities defined as increased signal intensity in >50% of the tibialis anterior muscle at MRI.
4. FEV1 and/or FVC < 60% of predicted.
5. Current or history of liver or renal disease.
6. Acute illness within 4 weeks prior to treatment (Day 1) which may interfere with the measurements.
7. Severe mental retardation which in the opinion of the investigator prohibits participation in this study.
8. Severe cardiac myopathy which in the opinion of the investigator prohibits participation in this study.
9. Need for mechanical ventilation.
10. Creatinine concentration above 1.5 times the upper limit of normal (age corrected).
11. Serum ASAT and/or ALAT concentration(s) which suggest hepatic impairment.
12. Use of anticoagulants, antithrombotics or antiplatelet agents.
13. Use of idebenone.
14. Use of any investigational product within 6 months prior to the start of the (pre)-screening for the study.
15. Subject has donated blood less than 90 days before the start of the (pre)-screening for the study.
16. Current or history of drug and/or alcohol abuse.
17. Participation in another trial with an investigational product.

Ages: 5 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-12; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Ferlini, PhD, Principal Investigator — Università di Ferrara and S.Anna Hospital, Ferrara, Italy; J. J. Verschuuren, MD, Principal Investigator — Leiden University Medical Center, Leiden, the Netherlands; N. Goemans, MD, Principal Investigator — UZ Leuven, Leuven, Belgium; M. Tulinius, MD, Principal Investigator — The Queen Silvia Children's Hospital, Gothenburg, Sweden
Locations (4):
- UZ Leuven, Leuven, Belgium
- S.Anna Hospital, Ferrara, Italy
- Leiden University Medical Center, Leiden, Netherlands
- The Queen Silvia Children's Hospital, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 Subjects were recruited to each of cohorts 1-6 (total n=18) for SC administration PRO044 9 of these 18 subjects were recruited to cohorts 7-9 (n=3 in each cohort) for IV adminstration PRO044
Pre-assignment Details: 3 Subjects were recruited to each of cohorts 1-6 (total n=18) for SC administration PRO044 9 of these 18 subjects were recruited to cohorts 7-9 (n=3 in each cohort) for IV adminstration PRO044
Groups:
- Subcutaneous PRO044 0.5 mg/kg: Subcutaneous injection of 0.5 mg/kg on day 1, 8, 15, 22 and 29.
  PRO044 SC: Subcutaneous injection, once a week, for five weeks
- Subcutaneous PRO044 1.5 mg/kg: Subcutaneous injection of maximally 1.5 mg/kg on day 1, 8, 15, 22 and 29.
  PRO044 SC: Subcutaneous injection, once a week, for five weeks
- Subcutaneous PRO044 5 mg/kg: Subcutaneous injection of maximally 5 mg/kg on day 1, 8, 15, 22 and 29.
  PRO044 SC: Subcutaneous injection, once a week, for five weeks
- Subcutaneous PRO044 8 mg/kg: Subcutaneous injection of maximally 8 mg/kg on day 1, 8, 15, 22 and 29.
  PRO044 SC: Subcutaneous injection, once a week, for five weeks
- Subcutaneous PRO044 10 mg/kg: Subcutaneous injection of maximally 10 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 SC: Subcutaneous injection, once a week, for five weeks
- Subcutaneous PRO044 12 mg/kg: Subcutaneous injection of maximally 12 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 SC: Subcutaneous injection, once a week, for five weeks
- Intravenous PRO044 1.5 mg/kg: Intravenous injection of maximally 1.5 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 IV: Intravenous injection, once a week, for five weeks
- Intravenous PRO044 5 mg/kg: Intravenous injection of maximally 5 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 IV: Intravenous injection, once a week, for five weeks
- Intravenous PRO044 8 mg/kg: Intravenous injection of maximally 8 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 IV: Intravenous injection, once a week, for five weeks
Period: Subcutaneous Cohort 1 - 6
Arm/Group | Subcutaneous PRO044 0.5 mg/kg | Subcutaneous PRO044 1.5 mg/kg | Subcutaneous PRO044 5 mg/kg | Subcutaneous PRO044 8 mg/kg | Subcutaneous PRO044 10 mg/kg | Subcutaneous PRO044 12 mg/kg | Intravenous PRO044 1.5 mg/kg | Intravenous PRO044 5 mg/kg | Intravenous PRO044 8 mg/kg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intravenous Period 7 - 9
Arm/Group | Subcutaneous PRO044 0.5 mg/kg | Subcutaneous PRO044 1.5 mg/kg | Subcutaneous PRO044 5 mg/kg | Subcutaneous PRO044 8 mg/kg | Subcutaneous PRO044 10 mg/kg | Subcutaneous PRO044 12 mg/kg | Intravenous PRO044 1.5 mg/kg | Intravenous PRO044 5 mg/kg | Intravenous PRO044 8 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO044, Cohort 1 | PRO044, Cohort 2 | PRO044, Cohort 3 | PRO044, Cohort 4 | PRO044, Cohort 5 | PRO044, Cohort 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 3 | 3 | 3 | 3 | 18
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 18
Region of Enrollment [Number; unit: participants]
  Belgium | 3 | 1 | 0 | 0 | 1 | 1 | 6
  Netherlands | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Italy | 0 | 0 | 3 | 1 | 1 | 2 | 7
  Sweden | 0 | 2 | 0 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Increase in Dystrophin Expression in the Muscle Biopsies by Immunofluorescence Analyses of Cross-sections and by Western Blot Analyses of Total Protein Extracts
Time Frame: Within 13 weeks after 5 weeks of treatment
Population: For some participants it was not possible to determine dystrophin expression in muscle biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | PRO044, Cohort 1 | PRO044, Cohort 2 | PRO044, Cohort 3 | PRO044, Cohort 4 | PRO044, Cohort 5 | PRO044, Cohort 6 | PRO044, Cohort 7 | PRO044, Cohort 8 | PRO044, Cohort 9
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 3 | 2 | 3 | 3
Participants | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 3 | 1

2. Primary Outcome: Safety and Tolerability of PRO044
Description: number of subjects with 1 or more treatment emergent adverse events following SC or IV PRO044
Time Frame: During the 5 weeks of treatment and during the 13 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PRO044, Cohort 1 | PRO044, Cohort 2 | PRO044, Cohort 3 | PRO044, Cohort 4 | PRO044, Cohort 5 | PRO044, Cohort 6 | PRO044, Cohort 7 | PRO044, Cohort 8 | PRO044, Cohort 9
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3

3. Secondary Outcome: PRO044 Pharmacokinetic Cmax (μg/mL) Following Subcutaneous Administration
Description: Pharmacokinetic population evaluated for maximum plasma concentration (Cmax)
Time Frame: Week 1, Week 5
Population: Pharmacokinetic population evaluated
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- PRO044, Cohort 7: IV injection of maximally 1.5 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 SC: IV, once a week, for five weeks
- PRO044, Cohort 8: IV injection of maximally 5 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 SC: IV, once a week, for five weeks
- PRO044, Cohort 9: IV injection of maximally 12 mg/kg on day 1, 8, 15, 22 and 29
  PRO044 SC: IV, once a week, for five weeks
Arm/Group | PRO044, Cohort 1 | PRO044, Cohort 2 | PRO044, Cohort 3 | PRO044, Cohort 4 | PRO044, Cohort 5 | PRO044, Cohort 6 | PRO044, Cohort 7 | PRO044, Cohort 8 | PRO044, Cohort 9
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
ug/mL
  Week 1 | 0.4 (42.5) | 1.6 (21.7) | 4.2 (61.5) | 6.2 (53.8) | 4.9 (21.7) | 5.2 (16.0) | 3.1 (28.9) | 4.7 (18.9) | 8.7 (31.3)
  Week 5 | 0.4 (28.8) | 1.5 (22.9) | 3.4 (31.4) | 5.1 (24.2) | 4.4 (7.0) | 4.8 (35.7) | 2.2 (20.6) | 3.5 (69.5) | 8.7 (33.6)

ADVERSE EVENTS:
Arm/Group | PRO044, Cohort 1 | PRO044, Cohort 2 | PRO044, Cohort 3 | PRO044, Cohort 4 | PRO044, Cohort 5 | PRO044, Cohort 6 | PRO044, Cohort 7 | PRO044, Cohort 8 | PRO044, Cohort 9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 2/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO044, Cohort 1 (N=3) | PRO044, Cohort 2 (N=3) | PRO044, Cohort 3 (N=3) | PRO044, Cohort 4 (N=3) | PRO044, Cohort 5 (N=3) | PRO044, Cohort 6 (N=3) | PRO044, Cohort 7 (N=3) | PRO044, Cohort 8 (N=3) | PRO044, Cohort 9 (N=3)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — fell over in playground
International normalised ratio increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
orthostatic proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRO044, Cohort 1 (N=3) | PRO044, Cohort 2 (N=3) | PRO044, Cohort 3 (N=3) | PRO044, Cohort 4 (N=3) | PRO044, Cohort 5 (N=3) | PRO044, Cohort 6 (N=3) | PRO044, Cohort 7 (N=3) | PRO044, Cohort 8 (N=3) | PRO044, Cohort 9 (N=3)
Injection site hematoma (General disorders) | 1 | 3 | 3 | 3 | 3 | 3 | 1 | 1 | 0
Injection site erythema (General disorders) | 0 | 3 | 3 | 3 | 2 | 3 | 0 | 2 | 0
Injection site edema (General disorders) | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site erythema (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Injection site discoloration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Edema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hookworm infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural edema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Complement factor decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
aPTT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Monocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RBC urine positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laboratory test abnormal (elevated MCP-1 levels) (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Complement factor C3 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystatin C increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GLDH increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
WBC count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoglobinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less